CLINICAL TRIAL: NCT06480942
Title: The Performance of Changes of Pulse Pressure and of Pulse Pressure Variation to Detect Preload Responsiveness in Spontaneously Breathing Patients
Brief Title: Arterial Pressure Derived Dynamic Parameters to Detect Preload Responsiveness in Spontaneously Breathing Patients
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO24013
Record Dates: First submitted 2024-06-10; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Hypovolemia
Keywords: Pulse Pressure; Pulse Pressure Variation; Passive Leg Raising; Echocardiography; Preload dependency
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive PLR test (PLR +): * Patient over 18 years old.
  * Hospitalized in intensive care.
  * For which the clinician in charge of the patient will need to predict the response to fluids and decide on a possible infusion of fluids, because of:
    * Acute circulatory failure with mean arterial pressure < 65mmHg or < 30mmHg of its baseline value for hypertensive patients.
    * And/or other signs of hemodynamic instability (tachycardia, mottling, oliguria, hyperlactatemia) :
  * In spontaneous ventilation and without ventilatory assistance.
  * Previously equipped with an arterial catheter.
  Interventions: Other: Detection of preload responders by a PLR test
- Negative PLR test (PLR-): * Patient over 18 years old.
  * Hospitalized in intensive care.
  * For which the clinician in charge of the patient will need to predict the response to fluids and decide on a possible infusion of fluids, because of:
    * Acute circulatory failure with mean arterial pressure < 65mmHg or < 30mmHg of its baseline value for hypertensive patients.
    * And/or other signs of hemodynamic instability (tachycardia, mottling, oliguria, hyperlactatemia) :
  * In spontaneous ventilation and without ventilatory assistance.
  * Previously equipped with an arterial catheter.
  Interventions: Other: Detection of preload responders by a PLR test

INTERVENTIONS:
Other: Detection of preload responders by a PLR test — Detection of preload dependency by using PLR test and echocardiography

SUMMARY:
The management of septic shock patients includes the infusion of fluids, however fluids may be deleterious if the patient does not respond by increasing cardiac output. By consequence, it is now recommended to predict the fluid response (fluid or preload responsiveness) before infusing them. In this protocol, the investigators will include critically ill patients spontaneously breathing, for whom the physician in charge has decided to test preload responsiveness. The investigators will collect from the continuous monitoring of arterial pressure of the patient the pulse pressure(PP) which is the difference between systolic arterial pressure and diastolic arterial pressure and the pulse pressure variation (PPV) automatically displayed by the monitor in addition to other clinical (hemodynamic, respiratory) parameters. After one minute of passive leg raising manoeuvre (PLR) the investigators collect the same parameters and the investigators will compare the changes of these parameters in patients who are preload responsive to patients who are not. Preload responsiveness will de defined by echocardiographic parameters before and during PLR. More exactly, a surrogate of cardiac output measured by echocardiography wich is VTI of the sub-aorti flow; an increase of more than 12% defines apreload responsive patient.

DETAILED DESCRIPTION:
*Objectives:

Primary : to assess the diagnostic performance of the decrease in pulse pressure variation (PPV) during a passive leg raising test (PLR) to predict preload responsiveness in spontaneously breathing patients hospitalized in intensive care.

Secondary:

* Evaluate the diagnostic performance of the increase in pulse pressure (PP) during a PLR test to predict preload responsiveness in this same population.
* Compare before/after PLR measurements other hemodynamic data (blood pressure, cardiac output, heart rate).

  * Experimental scheme: it is a diagnostic and monocentric study.
  * Population / patients:

Inclusion criteria:

* Patient over 18 years old.
* Hospitalized in intensive care.
* For which the clinician in charge of the patient will need to predict the response to fluids and decide on a possible infusion of fluids, because of:

  * Acute circulatory failure with mean arterial pressure < 65mmHg or < 30mmHg of its baseline value for hypertensive patients.
  * And/or other signs of hemodynamic instability (tachycardia, mottling, oliguria, hyperlactatemia).
* In spontaneous ventilation and without ventilatory assistance.
* Previously equipped with an arterial catheter.
* Affiliated to a social security scheme.

Non-inclusion criteria:

* Patient with arrythmia (PPV is not applicable).
* Patient with intra-abdominal hypertension (PLR test is not valid).
* Patient with a contraindication/impossibility to the PLR maneuver (lower limb amputation, respiratory intolerance).
* Patient with poor echogenicity noted previously.
* Patient protected by law.

  * Investigation Plan:

Patients meeting the inclusion criteria and not presenting any non-inclusion criteria may be included. The patient will be informed, or his/her relatives if he/she is unable to express their will, of the objectives and the progress of the study. If the patient, or his/her relatives, does not object to participate to the study, the course of the study will be as follows:

1. The following measurements will be performed before and after the PLR test in spontaneously breathing patients (SB) to evaluate the preload dependency:

   * Hemodynamic data: systolic (SAP), diastolic (DAP), mean (MAP), pulse pressure (PP), heart rate (HR), value of the Pulse Pressure Variation (PPV), cardiac index (CI) if cardiac output monitoring is already present.
   * Echographic data including: time-velocity integral of sub-aortic flow VTI Sub AO); aortic outflow chamber diameter (Diam outflow tract); data from the transmitral pulsed Doppler as well as the data from the tissue Doppler at the mitral annulus (E wave velocity; A wave; E' wave); left ventricular end-diastolic surface.
2. Collection of demographic parameters (age, sex, comorbidities), acute pathology and severity scores (SAPSII, APACHE II, SOFA) in the patient file.
3. Collection of oxygenation parameters: mode (conventional oxygen therapy or High Flow), Fio2 or liter O2/min, Flow if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Hospitalized in intensive care.
* For which the clinician in charge of the patient will need to predict the response to fluids and decide on a possible infusion of fluids, because of:

  * Acute circulatory failure with mean arterial pressure < 65mmHg or < 30mmHg of its baseline value for hypertensive patients.
  * And/or other signs of hemodynamic instability (tachycardia, mottling, oliguria, hyperlactatemia) :
* In spontaneous ventilation and without ventilatory assistance.
* Previously equipped with an arterial catheter.
* Affiliated to a social security scheme.

Exclusion Criteria:

* Patient with arrythmia (PPV is not applicable).
* Patient with intra-abdominal hypertension (PLR test is not valid).
* Patient with a contraindication/impossibility to the PLR maneuver (lower limb amputation, respiratory intolerance).
* Patient with poor echogenicity noted previously.
* Patient protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patient over 18 years old.
  * Hospitalized in intensive care.
  * For which the clinician in charge of the patient will need to predict the response to fluids and decide on a possible infusion of fluids, because of:
    * Acute circulatory failure with mean arterial pressure < 65mmHg or < 30mmHg of its baseline value for hypertensive patients.
    * And/or other signs of hemodynamic instability (tachycardia, mottling, oliguria, hyperlactatemia) :
  * In spontaneous ventilation and without ventilatory assistance.
  * Previously equipped with an arterial catheter.
  * Affiliated to a social security scheme.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the decrease in Pulse Pressure Variation (PPV) during a Passive Leg Raising test (PLR) to predict preload responsiveness | Day 1
  To assess the diagnostic performance of the decrease in pulse pressure variation (PPV) during a passive leg raising test (PLR) to predict preload responsiveness in spontaneously breathing patients hospitalized in intensive care.

SECONDARY OUTCOMES:
Evaluate the diagnostic performance of the increase in pulse pressure (PP) during a PLR test to predict preload responsiveness | Day 1
  Evaluate the diagnostic performance of the increase in pulse pressure (PP) during a PLR test to predict preload responsiveness in spontaneously breathing patients hospitalized in intensive care.
Compare PLR measurements other hemodynamic data | Day 1
  Compare before/after PLR measurements other hemodynamic data in spontaneously breathing patients hospitalized in intensive care.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Background] Shi R, Moretto F, Prat D, Jacobs F, Teboul JL, Hamzaoui O. Dynamic changes of pulse pressure but not of pulse pressure variation during passive leg raising predict preload responsiveness in critically ill patients with spontaneous breathing activity. J Crit Care. 2022 Dec;72:154141. doi: 10.1016/j.jcrc.2022.154141. Epub 2022 Sep 15. PMID 36116288
- [Background] Hamzaoui O, Shi R, Carelli S, Sztrymf B, Prat D, Jacobs F, Monnet X, Gouezel C, Teboul JL. Changes in pulse pressure variation to assess preload responsiveness in mechanically ventilated patients with spontaneous breathing activity: an observational study. Br J Anaesth. 2021 Oct;127(4):532-538. doi: 10.1016/j.bja.2021.05.034. Epub 2021 Jul 8. PMID 34246460